CLINICAL TRIAL: NCT02210260
Title: Pain Relief After Colorectal Surgery: Single-shot Spinal Combined With Painbuster® vs Painbuster® Alone. A Pilot Randomised Controlled Trial
Brief Title: Pain Relief After Colorectal Surgery: Spinal Combined With Painbuster® vs Painbuster® Alone.
Acronym: PROSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNE 2190
Record Dates: First submitted 2014-07-31; First posted 2014-08-06 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: Cancer; Colorectal; Pain relief
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Bupivacaine; Heroin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous infusion of local anaesthetic (Active Comparator): Continuous infusion of local anaesthetic into the surgical wound
  Interventions: Procedure: Continuous infusion of local anaesthetic; Drug: Bupivacaine; Device: A Painbuster® catheter
- Spinal and infusion of local anaesthetic (Experimental): A one off spinal anaesthetic plus a continuous infusion of local anaesthetic into the surgical wound
  Interventions: Procedure: Spinal and infusion of local anaesthetic; Drug: Bupivacaine; Drug: Diamorphine; Device: A Painbuster® catheter; Device: 25G Whitacre needle

INTERVENTIONS:
Procedure: Spinal and infusion of local anaesthetic — Spinal anaesthetic will be performed in the lateral position using a midline approach. L3/4 interspace will be identified using Tuffier's as the anatomical landmark. After confirmation of correct placement using a 25G Whitacre needle, 12.5 mg of hyperbaric Bupivacaine in a mixture with 500mcg Diamorphine will be injected intrathecally.
  PLUS
  Painbuster® catheters will be placed by the surgeon at the end of the procedure in a location determined by the surgical approach. A bolus dose of 20ml 0.25% L-Bupivacaine will be injected down the catheters prior to the connection of the elastomeric pump which will also contain 270ml 0.25% L-Bupivacaine.
  Arms: Spinal and infusion of local anaesthetic
Procedure: Continuous infusion of local anaesthetic — A Painbuster® catheter will be placed by the surgeon at the end of the procedure in a location determined by the surgical approach. A bolus dose of 20ml 0.25% L-Bupivacaine will be injected down the catheters prior to the connection of the elastomeric pump which will also contain 270ml 0.25% L-Bupivacaine.
  Arms: Continuous infusion of local anaesthetic
Drug: Bupivacaine
Drug: Diamorphine — 500mcg
  Arms: Spinal and infusion of local anaesthetic
Device: A Painbuster® catheter
Device: 25G Whitacre needle
  Arms: Spinal and infusion of local anaesthetic

SUMMARY:
Limiting surgical stress and managing postoperative pain are well understood to influence recovery and outcome from major surgery for colorectal cancer and both are fundamental aspects of enhanced recovery protocols.

Traditional approaches for dealing with these problems such as epidural or patient controlled intravenous opioid analgesia are associated with problems that may be detrimental to postoperative recovery and surgical outcome. As a result there is evidence in the literature of increasing interest in alternative techniques such as intrathecal anaesthesia or continuous wound infusion of local anaesthetic, however nobody has examined the effect of combining the techniques or their impact on the surgical stress response.

We intend to compare patients undergoing major resections for colorectal cancer receiving intrathecal anaesthesia in combination with a wound infusion of local anaesthetic with those receiving a continuous wound infusion alone. We will examine the surgical stress response and postoperative pain control in addition to objective measures of postoperative recovery.

We suggest that our approach will attenuate the surgical stress response and provide optimal pain control that will ultimately translate in improved recovery and outcome following surgery for colorectal cancer.

DETAILED DESCRIPTION:
This is a pilot randomised controlled trial

Hypotheses -

Following colorectal surgery, spinal anaesthesia combined with a continuous infusion of local anaesthetic into the surgical wound provides

1. better pain relief
2. a reduced stress response

when compared to the use of continuous infusion of local anaesthetic into the surgical wound alone.

Patients undergoing surgical resection for colorectal cancer will be randomised to receive either

1. A single shot of spinal anaesthesia plus a continuous infusion of local anaesthetic into the surgical wound or
2. Continuous infusion of local anaesthetic into the surgical wound

Spinal Anaesthesia

The spinal anaesthetic (SA) with be placed after commencement of general anaesthesia this will ensure the patients remain blinded to the intervention. SA will be performed in the lateral position using a midline approach. L3/4 interspace will be identified using Tuffier's as the anatomical landmark. After confirmation of correct placement using a 25G Whitacre needle, 12.5 mg of hyperbaric Bupivacaine in a mixture with 500mcg Diamorphine will be injected intrathecally.

Infusion of local anaesthetic

The catheter through which the infusion of local anaesthetic will be given, will be placed by the surgeon at the end of the procedure in a location determined by the surgical approach. A bolus dose of 20ml 0.25% L-Bupivacaine will be injected down the catheters prior to the connection of the elastomeric pump which will also contain 270ml 0.25% L-Bupivacaine

General anaesthesia will be managed in the same way for both groups

ELIGIBILITY:
Inclusion Criteria:

* All patients who are undergoing either laparoscopic or open colorectal resections will be considered eligible for the study.

Exclusion Criteria:

* Patients under 18 years of age.
* Pregnant females.
* Patients undergoing an abdominoperineal resection.
* Patients who will not contemplate being randomized to receive a spinal anaesthetic.
* Patients with a history of failure to place an epidural / spinal anaesthetic.
* Hypersensitivity to local anaesthetics.
* Lack of capacity to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Neuroendocrine response to surgery | 24 hours
  Peripheral blood samples taken at baseline, 60 minutes after surgical incision and 24 hours postoperatively will be analysed for cortisol and noradrenaline.

SECONDARY OUTCOMES:
Length of hospital stay or fitness for discharge | Up to 12 days
  Discharge criteria:
  1. Good pain control with oral analgesia.
  2. Tolerating solid food without nausea and vomiting.
  3. No IV fluid or medication.
  4. Independently mobile and self-caring or at the same level as prior to admission.
  5. Stable observations and blood biochemistry.
  6. No other concerns or complications preventing discharge.
Postoperative complications | Up to 12 days
  All complications in the postoperative period will be recorded. Particular emphasis will be given to:
  Wound infection
  Cardiac failure:
  Complications related to spinal anaesthesia.
  Adequacy of deep vein thrombosis prophylaxis.
Episodes of hypotension in the postoperative period | Up to 12 days
  This will be defined as a sustained systolic blood pressure of less than 90 mm/Hg.
Postoperative pain | Up to 72 hours after surgery
  This will be assessed using a visual analogue scale . Measurements will be taken in recovery then once a day for 72 hours postoperatively. Pain scores will be measured at rest and on coughing.
Postoperative analgesic requirement | Up to 72 hours after surgery
  The total quantity and type (opiate or non-opiate) of all analgesics administered for 72 hours postoperatively.
Amount of postoperative IV fluid administered | Up to 12 days
  Total amount of IV fluid given in postoperative period
Postoperative mobility | Up to 12 days
  Postoperative mobility will be assessed as
  time until able to stand aided and unaided,
  duration of time spent out of bed on each postoperative day
  maximum walking distance with assistance on a daily basis.
Return of gut function | Up to 12 days
  4.2.8 Time to return of gut function This is defined by the oral/enteral tolerance of > 80% of nutritional requirement.
  These requirements will be assessed individually for each patient in the study by an appropriately trained dietician
Oxidative stress | For 24 hours
  Peripheral blood samples will be taken at baseline, 60 minutes after surgical incision and 24 hours postoperatively and analysed for heat shock proteins 37 and 32.
Inflammatory pathway | Up to 24 hours after surgery
  Peripheral blood samples taken at baseline, 60 minutes after surgical incision and 24 hours postoperatively will be analysed for IL1.
  Peritoneal biopsies taken prior to closure of surgical wound and analysed for IL1.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Harper, MBChB, FRCA, Principal Investigator — York Teaching Hospital NHS Foundation Trust
Locations (1):
- Scarborough General Hospital, Scarborough, North Yorkshire, United Kingdom